CLINICAL TRIAL: NCT05095181
Title: Preventive and Personalized Medicine (2021-2023)
Brief Title: To Study the Effects of Host Genetic Factors on Liver Cirrhosis
Status: Completed | Type: Observational
Sponsor: Asfendiyarov Kazakh National Medical University (Other)
Responsible Party: Principal Investigator, Ildar Fakhradiyev, Head of the Laboratory of Experimental Medicine, Asfendiyarov Kazakh National Medical University
Other Study IDs: 1188
Record Dates: First submitted 2021-10-21; First posted 2021-10-27 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Liver Cirrhosis
Keywords: SNP
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group:: patients with liver cirrhosis
  Interventions: Genetic: SNP analysis of the DNA
- Control group: patients without liver cirrhosis
  Interventions: Genetic: SNP analysis of the DNA

INTERVENTIONS:
Genetic: SNP analysis of the DNA — SNP analysis of the DNA obtained from peripheral blood sample

SUMMARY:
The purpose of this study is to identify genetic determinants of susceptibility to liver cirrhosis . It will assist in predicting individual risks of disease progression and would help to clarify pathophysiologic mechanisms of liver cirrhosis .

ELIGIBILITY:
Inclusion Criteria:

* hepatitis B

Exclusion Criteria:

* the casual aget of liver disease is not viral infection, such as alcohol abuse

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: KAZAKH POPULATION
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
genotyping for the SNP associated with liver cirrhosis | 1 year
  Genotype frequency of SNP in the study genes of participants and control participants.

CONTACTS AND LOCATIONS:
Overall Officials: Bibigul Saparbekovna, PhD, Principal Investigator — JSC "National Scientific Center of Surgery named after A.N. Syzganova "
Locations (1):
- National Scientific Center of Surgery named after A.N. Syzganova, Almaty, Kazakhstan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ilyassova BS, Abzhaparova B, Smailova DS, Bolatov A, Baymakhanov B, Beloussov V, Solomadin M, Shamsivaliyeva K, Alpysbayava G, Issakova G, Granica J, Mukushkina D, Sagatov IY, Kaniyev S. Prevalence and genotypes distribution of virus hepatitis B and hepatitis delta virus in chronic liver diseases in Kazakhstan. BMC Infect Dis. 2023 Aug 14;23(1):533. doi: 10.1186/s12879-023-08524-1. PMID 37580657